CLINICAL TRIAL: NCT06763380
Title: Comparison of Ultrasound and Hysterosalpingography in Evaluation of Uterine Abnormality in Patients With Primary and Secondary Infertility
Brief Title: Comparison of Ultrasound and Hysterosalpingography in Evaluation of Uterine Abnormality in Patients With Infertility
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/012
Record Dates: First submitted 2024-12-17; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Uterine Abnormality
MeSH Terms: conditions — Uterine Anomalies | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — Detection of uterine abnormalities in patients who are infertile buy using Ultrasound
Diagnostic Test: ultrasound then hysterosalpingography — If uterine abnormality could not diagnosed with ultrasound then hysterosalpingography would be performed

SUMMARY:
The leading issue that every couple is experiencing in present era is infertility and it has become the major problem worldwide. Many hormonal disorders, weight, diet, and uterine abnormalities contributes in infertility.

DETAILED DESCRIPTION:
To Compare diagnostic effectiveness of Ultrasound and Hysterosalpingography in detecting uterine abnormalities among Primary and Secondary Infertile women.

In order to obtain the necessary results, 73 patients were examined on Ultrasound and then referred for Hysterosalpingography at Radiology Department of Dr.Essa Lab and Punjab Radiology. Patients with Primary and secondary infertility between the age of 18 to 45 were included whereas pregnant women and women with PID and GTI were excluded. The data were collected utilizing the questionnaire and then processed in SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* primary and secondary infertile women

Exclusion Criteria:

* Pregnant women. Women with PID

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Infertility
Study Population: primary and secondary infertile women using Ultrasound and Hysterosalpingography in Evaluation of Uterine Abnormality
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
2D Ultrasound Scan | 12 Months
  Uterine anomalies can be diagnosed on routine two-dimensional ultrasound scan
Hysterosalpingography test | 12 Months
  HSG is an x-ray exam of the uterus and fallopian tubes. It uses a special form of x-ray called fluoroscopy and a contrast materia.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Essa Lab, High Q tower, Jail Road Lahore", Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No